CLINICAL TRIAL: NCT00981370
Title: Clinical Importance of Treating Iron Overload in Sickle Cell Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: 1 consented patient never started on study drug, lost to follow up
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Thomas Coates, Division Head of Hematology, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670AUS30T
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Anemia, Sickle Cell; Transfusion Hemosiderosis
Keywords: Sickle Cell Disease; Sickle Cell Anemia; Iron Overload; Chelation Therapy; Iron overload from blood transfusions; Heart rate variability; Autonomic dysfunction
MeSH Terms: conditions — Anemia, Sickle Cell; Iron Overload; Primary Dysautonomias | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm study (Other): Single Arm study, all subjects to receive study medication, deferasirox (Exjade).
  Interventions: Drug: deferasirox

INTERVENTIONS:
Drug: deferasirox — Treatment starting dose of 20mg/kg/day based on subjects baseline LIC (liver iron concentration) and gradually escalate the dose to a maximum of 35 mg/kg/day based upon toxicity. Duration is up to a max of 12 months.
  Other Names: Exjade

SUMMARY:
Hypothesis:

The investigators suspect that significant degrees of iron overload in subjects with SCD result in decreased red cell survival, abnormal endothelial function and markedly dysregulated autonomic function. Furthermore, the investigators anticipate that the magnitude of these effects is proportional not only to the magnitude of total body iron stores but also to the duration of exposure to the high iron levels in tissues.

Primary objective To determine if red cell survival as assessed by 51Cr red cell survival analysis, hemoglobin level, reticulocyte count, lactic acid dehydrogenase, and plasma hemoglobin in sickle cell patients is related to the degree of iron overload.

Secondary objective(s)

1. Determine if the magnitude of endothelial-dependant vasodilation is related to The degree of iron overload.
2. Determine if the degree of change in cardiac beat to beat variability in response to hypoxic exposure or to cold exposure ("cold-face-test") is related the magnitude of iron overload.

The primary measure of iron overload will be MRI determination of liver iron concentration.

DETAILED DESCRIPTION:
Patients with sickle cell anemia often require blood transfusion as part of the treatment for their disease. Since each teaspoon of packed red blood cells contains about 5 mg of iron and humans have no way to get rid of excess iron, the levels of iron in sickle cell patients increase rapidly with each transfusion. Too much iron is extremely dangerous and causes damage to blood vessels, red blood cells, liver, hormone producing glands and heart. It is very difficult to know what damage due to iron overload in sickle cell patients because the sickle cell disease itself causes organ damage to the same organs affected by iron.

The purpose of this project is to demonstrate that iron overload significantly increases the morbidity of sickle cell disease and that treatment of the iron overload with Exjade® prevents or attenuates iron-related morbidity. To accomplish this we will screen sickle cell patients with a history of many blood transfusions to see if they have high iron levels. Then we will treat the patients who have very high iron levels with a drug which will remove the iron. Only patients with a very high iron level will be eligible for the treatment. These patients will have been transfused many times before but cannot currently be on blood transfusions. Before we start the treatment we will test the level of anemia, how fast the red cells are being destroyed, how well their blood vessels work and how well their heart works. When the treatment is over, we will repeat these tests and see if there is an improvement.

To qualify for this study, you must carry the diagnosis of sickle cell anemia and you must have received 10 or more blood transfusions in your life. You also cannot currently be on a regular transfusion program where you are getting blood transfusions regularly planned more than three times a year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with sickle cell anemia (SS or SB thalassemia) with transfusional iron overload.
* Currently not on chronic or frequent transfusion
* Age equal or greater then 14 years
* Patients with iron overload from repeated blood transfusion, as defined by one of the following:

  1. For patients greater then 16 years old receiving simple transfusions: estimated lifetime history of receipt of at least 100 ml/kg or 15 adult units of packed red blood cells, OR
  2. For patients equal to or less then 16 years old receiving simple transfusions: estimated lifetime history of receipt of at least 100 ml/kg of packed red blood cells, OR
  3. For any patient: liver iron content equal/greater then 3 mg Fe/g dw as measured by biopsy or magnetic resonance imaging who have not been adequately chelated since that measurement, OR
  4. a serum ferritin equal/greater then 1000 ng/mL on at least two occasions, at least two weeks apart, during the prior year. Samples must be obtained in the absence of concomitant infection
* Life expectancy equal/greater then 12 months
* Sexually active women must use an effective method of contraception, or must have undergone clinically documented total hysterectomy and/or oophorectomy, or tubal ligation or be postmenopausal (defined as amenorrhea for at least 12 months)

Inclusion criteria for treatment pilot study

* Meets all inclusion criteria for screening
* LIC by MRI greater than or equal to 8 mg/g.

Exclusion Criteria:

* Blood transfusion within 12 weeks of the day 0 hemolysis labs
* Currently requires blood transfusion more than three times a year.
* Contraindication to MRI, including cardiac pacemaker, brain aneurysm clip, implanted neurostimulator, insulin pump, cochlear implant, metal slivers in the eyes, intrauterine device or any other MRI incompatible metal implants or intractable claustrophobia.
* Serum creatinine above the upper limit of normal
* Concomitant treatment with erythropoietin or its analogs.
* AST or ALT greater then 250 U/L during screening (patients may be re-screened at a later date if the cause of the elevation is known to be due to a transient process).
* Patients receiving currently on chelation will be asked to stop for one week before starting or restarting Exjade. (a equal/greater then 1 week washout period prior to first dose of study drug is required)
* History of HIV positive test result (ELISA or Western blot)
* History of drug or alcohol abuse within the 12 months prior to enrollment
* Patients with uncontrolled systemic hypertension
* Severe cardiac insufficiency (NYHA III or IV), with uncontrolled and/or unstable cardiac or coronary artery disease not controlled by standard medical therapy
* Patients with a diagnosis of or history of clinically relevant ocular toxicity related to iron chelation
* Systemic diseases (cardiovascular, renal, hepatic, etc.) which would prevent study treatment
* Pregnancy (as documented in required screening laboratory test) or breast feeding
* Patients who received treatment with systemic investigational drug within the past 4 weeks or topical investigational drug within the past 7 days or are planning to receive other investigational drugs while participating in the study
* Other surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of study drug
* History of non-compliance to medical regimens or patients who are considered potentially unreliable and/or not cooperative

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D. Coates, M.D., Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Childrens Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
no data entered, no subjects enrolled

REFERENCES:
- [Background] Cappellini MD, Cohen A, Piga A, Bejaoui M, Perrotta S, Agaoglu L, Aydinok Y, Kattamis A, Kilinc Y, Porter J, Capra M, Galanello R, Fattoum S, Drelichman G, Magnano C, Verissimo M, Athanassiou-Metaxa M, Giardina P, Kourakli-Symeonidis A, Janka-Schaub G, Coates T, Vermylen C, Olivieri N, Thuret I, Opitz H, Ressayre-Djaffer C, Marks P, Alberti D. A phase 3 study of deferasirox (ICL670), a once-daily oral iron chelator, in patients with beta-thalassemia. Blood. 2006 May 1;107(9):3455-62. doi: 10.1182/blood-2005-08-3430. Epub 2005 Dec 13. PMID 16352812
- [Background] Vichinsky E, Onyekwere O, Porter J, Swerdlow P, Eckman J, Lane P, Files B, Hassell K, Kelly P, Wilson F, Bernaudin F, Forni GL, Okpala I, Ressayre-Djaffer C, Alberti D, Holland J, Marks P, Fung E, Fischer R, Mueller BU, Coates T; Deferasirox in Sickle Cell Investigators. A randomised comparison of deferasirox versus deferoxamine for the treatment of transfusional iron overload in sickle cell disease. Br J Haematol. 2007 Feb;136(3):501-8. doi: 10.1111/j.1365-2141.2006.06455.x. PMID 17233848
- [Background] Natta C, Creque L, Navarro C. Compartmentalization of iron in sickle cell anemia--an autopsy study. Am J Clin Pathol. 1985 Jan;83(1):76-8. doi: 10.1093/ajcp/83.1.76. PMID 3966442
- [Background] Koduri PR. Iron in sickle cell disease: a review why less is better. Am J Hematol. 2003 May;73(1):59-63. doi: 10.1002/ajh.10313. PMID 12701123
- [Background] Castro O, Poillon WN, Finke H, Massac E. Improvement of sickle cell anemia by iron-limited erythropoiesis. Am J Hematol. 1994 Oct;47(2):74-81. doi: 10.1002/ajh.2830470203. PMID 7522396
- [Background] Romero Mestre JC, Hernandez A, Agramonte O, Hernandez P. Cardiovascular autonomic dysfunction in sickle cell anemia: a possible risk factor for sudden death? Clin Auton Res. 1997 Jun;7(3):121-5. doi: 10.1007/BF02308838. PMID 9232355
- [Background] Wood JC, Ghugre N. Magnetic resonance imaging assessment of excess iron in thalassemia, sickle cell disease and other iron overload diseases. Hemoglobin. 2008;32(1-2):85-96. doi: 10.1080/03630260701699912. PMID 18274986
- [Background] Cheung YF, Chan GC, Ha SY. Arterial stiffness and endothelial function in patients with beta-thalassemia major. Circulation. 2002 Nov 12;106(20):2561-6. doi: 10.1161/01.cir.0000037225.92759.a7. PMID 12427652
- [Background] Sangkatumvong S, Khoo MC, Coates TD. Abnormal cardiac autonomic control in sickle cell disease following transient hypoxia. Annu Int Conf IEEE Eng Med Biol Soc. 2008;2008:1996-9. doi: 10.1109/IEMBS.2008.4649581. PMID 19163084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from local physicians and at CHLA.
Pre-assignment Details: No groups for this study.
Groups:
- Group One: No enrollment
Period: Overall Study
Arm/Group | Group One
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: First group of subjects to be enrolled.
Arm/Group | Group 1
Number analyzed (Participants) | 0
Age, Customized | 0
Gender
  Female | 0
  Male | 0
Liver Iron Concentration > 8mg/g dry weight | 0

OUTCOME MEASURES:

1. Primary Outcome: To Determine if Red Cell Survival as Assessed by Hemoglobin Level, Reticulocyte Count, Lactic Acid Dehydrogenase, and Plasma Hemoglobin in Sickle Cell Patients is Related to the Degree of Iron Overload
Time Frame: Baseline, 6 months and 12 months
Groups:
- Group 1: First group of subjects enrolled.
Arm/Group | Group 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was not collected. Only 1 subject passed screening to be enrolled but was then lost to follow up and never started study drug.
Groups:
- Group 1: No patients enrolled
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
1 consent patient, never treated, lost to follow up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No